CLINICAL TRIAL: NCT05190744
Title: A Multi-center, Open-Label, Exploratory Study to Assess the Efficacy of PB in Decreasing the Urine Output and Increasing the Urine Osmolality in Patients With Hereditary Nephrogenic Diabetes Insipidus, Patients With Autosomal Dominant Polycystic Kidney Disease Treated With Tolvaptan, And Severely Polyuric Patients With Previous Lithium Administration (Serendipity-PB1)
Brief Title: Probenecid (PB) to Treat Hereditary Nephrogenic Diabetes Insipidus (NDI), ADPKD Treated With Tolvaptan, and Severely Polyuric Patients With Previous Lithium Administration
Acronym: SerendipityPB1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Fouad T. Chebib, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-005437
Record Dates: First submitted 2021-12-29; First posted 2022-01-13 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease; Nephrogenic Diabetes Insipidus; Acquired Nephrogenic Diabetes Insipidus; Congenital Nephrogenic Diabetes Insipidus
Keywords: Tolvaptan; ADPKD; Polycystic Kidney Disease; Nephrogenic Diabetes Insipidus (NDI); Nephrogenic diabetes insipidus; Inherited nephrogenic diabetes insipidus; Diabetes Insipidus; Lithium; Lithium-induced nephrogenic diabetes insipidus; Vasopressin receptor antagonist; Tolvaptan-induced aquaresis
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Diabetes Insipidus, Nephrogenic; Polycystic Kidney Diseases; Diabetes Insipidus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Polyuric subjects with Hereditary Nephrogenic Diabetes Insipidus (Experimental): Polyuric subjects with hereditary nephrogenic diabetes insipidus with loss of function of arginine vasopressin receptor 2 (AVPR2) or aquaporin 2 (AQP2) will be treated with PB
  Interventions: Drug: PB
- Polyuric subjects with Autosomal Dominant Polycystic Kidney Disease treated with Tolvaptan (Experimental): Polyuric subjects with autosomal dominant polycystic kidney disease on chronic tolvaptan treatment will be treated with PB
  Interventions: Drug: PB
- Polyuric subject secondary to lithium administration (Experimental): Polyuric subject post lithium administration will receive PB
  Interventions: Drug: PB

INTERVENTIONS:
Drug: PB — 1000mg twice daily (BID). The dose of PB inducing the maximal increase in urine osmolality will be continued for up to four weeks providing that no side effects are observed including clinical and laboratory surveillance.

SUMMARY:
The purpose of this research is to study the effectiveness and safety of the medication PB in slowing the frequent urination related to tolvaptan as long-term treatment of Autosomal Dominant Polycystic Kidney Disease (ADPKD), or frequent urination related to inherited nephrogenic diabetes insipidus as an inherited condition or as an acquired condition from prior treatment with lithium.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥ 18 years of age (inclusive) at time of screening
* Diagnosis of one of the following:

  1. ADPKD(as delineated in cohort 1)
  2. Congenital NDI (as delineated in cohort 1)
  3. Lithium-induced NDI (as delineated in cohort 1)
* Glomerular filtration rate (GFR) ≥ 25 ml/min/1.73 m2 at time of screening visit calculated as in cohort
* 24 hours urine volume in baseline 1 visit ≥ 5000 ml/ day
* If hypertensive, blood pressure controlled on antihypertensives (<130/80 mm Hg) at least 30 days before day 1. Antihypertensives may be adjusted at time of baseline 2 per PI discretion.
* Female participants (see details in cohort 1 inclusion criteria)
* Have read, understood, and provided written informed consent after the nature of the study has been fully explained and must be willing to comply with protocol requirements and study-related procedures.
* Negative urinary pregnancy test (if applicable) at baseline 2
* Capable of providing urine samples as dictated by the protocol

Exclusion Criteria:

* Advanced diabetes (e.g., glycosylated hemoglobin [HgbA1c] >7.5%, and/or glycosuria by dipstick, significant proteinuria [>300 mcg albumin/mg creatinine]), other significant kidney disease, kidney cancer, transplanted kidney, single kidney, kidney surgery within the past 6 months (including cyst drainage or fenestration) or acute kidney injury within 6 months prior to screening.
* Clinically significant incontinence, overactive bladder, or urinary retention (e.g., benign prostatic hyperplasia).
* Other significant chronic medical disease (heart failure, diabetes mellitus, liver disease, transient or persistent elevated transaminases)
* History of acute gout attack in the past 30 days
* History of clinically significant drug or alcohol abuse in the 2 years prior to screening visit.
* Uncontrolled hyperuricemia or active gout
* History of hepatotoxicity related to tolvaptan; or clinically significant liver disease or impairment; or alanine aminotransferase (ALT), aspartate aminotransferase (AST), or total bilirubin values >1.2 x Upper Limit of Normal (ULN) during screening.
* Medical history or findings that preclude safe participation in the trial or participants who are likely to be non-compliant with trial procedures in the opinion of the investigator or medical monitor.
* Requirement for ongoing diuretic use.
* Participants who are currently taking, or are expected to be taking, strong or moderate CYP3A4 or CYP2C8 inhibitors or inducers including regular use of grapefruit juice, Seville oranges, or St. John's wort. If applicable, there should be a 14-day washout of these treatments prior to Day 1.
* Prior use of a sodium-glucose cotransporter 2 inhibitor (SGLT2i) (e.g., canagliflozin, dapagliflozin, empagliflozin, etc.) within the 2 months prior to screening visit or expected need for initiation of treatment with a SGLT2i inhibitor during the study. Current use of SGLT2i will be reviewed by PI and allow enrollment if patient has been on stable dose for at least 2 months.
* Prior use of a hypoxia-inducible factor prolyl hydroxylase (HIF-PH) inhibitor within the 2 months prior to screening visit or expected need for initiation of treatment with a HIF-PH inhibitor during the study;
* Participants who have taken any investigational drug or used an investigational device within 30 days, or 5 half-lives, whichever is longer, prior to screening visit 1a or plan to participate in an interventional trial during the study.
* Allergy to probenecid
* History of persistent hyponatremia
* Positive test results for hepatitis B surface antigen (HBsAg).
* Positive test results for hepatitis C (HCV) antibody (Anti-HCV), with the exception of participants for whom the reflex HCV RNA titer test is negative.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Change in urine osmolality | Baseline, 30 days
  Measured in milliosmoles per kilogram of water (mOsm/kg) from a urine specimen and is a measure of the concentration of osmotically active particles, principally sodium, chloride, potassium, and urea

SECONDARY OUTCOMES:
Change in urine output | From Baseline 2 to Post Treatment Follow Up at the end of 5 weeks
  Measured in milliliters per day (ml/day) by 24 hour urine collection

CONTACTS AND LOCATIONS:
Overall Officials: Fouad Chebib, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20525492